CLINICAL TRIAL: NCT00847808
Title: A Phase 3b Multicenter, Single-Blind Trial to Evaluate the Efficacy of Dexlansoprazole MR 30 mg in Maintaining Control of Gastroesophageal Reflux Disease Symptoms in Subjects on Prior Twice Daily Proton Pump Inhibitor Therapy
Brief Title: Efficacy of Dexlansoprazole MR on Heartburn Control in Participants Previously Receiving Twice Daily Proton Pump Inhibitor Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: T-GD08-178; U1111-1112-1761 (Registry Identifier: WHO)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Gastroesophageal Reflux
Keywords: Esophageal Reflux; Gastro-Esophageal Reflux; Gastroesophageal Reflux Disease; GERD; Regurgitation, Gastric; Heartburn; Drug Therapy
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngopharyngeal Reflux; Heartburn | interventions — Dexlansoprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dexlansoprazole MR QD

INTERVENTIONS:
Drug: Dexlansoprazole MR QD — Dexlansoprazole MR 30 mg, capsules and dexlansoprazole MR placebo-matching capsules, orally, each once daily for up to 6 weeks.
  Other Names: TAK-390; T-168390; TAK-390MR; Kapidex; Dexilant

SUMMARY:
The purpose of this study is to determine if patients with well-controlled heartburn symptoms on twice-daily proton pump inhibitor therapy remain well-controlled after stepping down to once-daily (QD) dexlansoprazole modified release (MR) 30 mg.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is recognized as a common and persistent medical problem in the US adult population. Gastroesophageal reflux disease comprises a spectrum of acid-related disorders including symptomatic nonerosive gastroesophageal reflux disease and erosive esophagitis. It affects men and women in nearly equal proportions, and the severity and intensity of heartburn symptoms may be similar in both types of patients.

Dexlansoprazole modified release is a dual delayed release formulation that consists of two types of granules contained in a single capsule. This dual delayed release formulation is designed to extend the duration of drug exposure and maintain pharmacologically active levels over a longer time period.

The purpose of this study is to demonstrate that participants with gastroesophageal reflux disease whose symptoms are well-controlled on twice daily proton pump inhibitors, remain well-controlled when switched to dexlansoprazole MR.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to any study-specific procedures being performed, the participant voluntarily signs an Investigational Review Board-approved informed consent form (ICF) and any privacy statement/authorization form required (eg, The Health Insurance Portability and Accountability Act (HIPAA) authorization)
2. Has a history of gastroesophageal reflux disease symptom, including heartburn, prior to therapy, who are currently being treated with twice daily proton pump inhibitors, excluding Dexilant (dexlansoprazole).
3. Taking a stable dose of any twice daily proton pump inhibitors for less than or equal to 1 year and greater than 8 weeks prior to Screening.
4. Participant is well-controlled on their current twice daily proton pump inhibitors.
5. Females cannot be nursing and must have a negative urine pregnancy test at Day -1 or be of non-childbearing potential. If females are of child bearing potential, must have a negative serum human chorionic gonadotropin (hCG) pregnancy test during Screening and on an acceptable form of contraception, or have had bilateral tubal ligation if performed a minimum of 90 days prior to Day 1.

Exclusion Criteria:

1. Has a history of co-existing diseases affecting the esophagus, history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
2. Has active gastric or duodenal ulcers during the 30 days prior to Screening.
3. Has acute upper gastrointestinal hemorrhage during the 30 days prior to Screening.
4. Has current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition.
5. Has known hypersensitivity to any proton pump inhibitor or any component of dexlansoprazole MR.
6. Use of any Histamine type-2 receptor antagonist or antacids during Screening or anticipated use during the study treatment period.
7. Use of the following medications 7 days prior to Screening or anticipated use during the study:

   * Sucralfate.
   * Misoprostol.
   * Systemic corticosteroids.
   * Prokinetics (to include metoclopramide, cisapride, tegaserod).
   * Bisphosphonates during the 6 months prior to Screening or anticipated use during the study.
   * Chronic use (> 12 doses per month) of nonsteroidal anti-inflammatory drugs
   * Drugs with significant anticholinergic effects such as tricyclic antidepressants or drugs with central nervous system effects that could mask perception of symptoms.
   * Any investigational drug(s) within 30 days of Screening.
8. Has received blood products within the 3 months prior to Screening.
9. History of alcohol abuse or illegal drug use or drug addiction in the 12 months prior to Screening.
10. Evidence of uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
11. Atypical manifestations of gastroesophageal reflux disease.
12. Has abnormal screening laboratory values that suggest a clinically significant underlying disease or condition.
13. Cancer within 5 years prior to Screening.
14. Is known to have acquired immunodeficiency syndrome.
15. Has any condition that is likely to require inpatient surgery during the course of the study.
16. Surgery of the acute upper gastrointestinal tract, including bariatric.
17. Is in the opinion of the investigator unable to comply with the requirements of the study or are unsuitable for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (52):
- United States (52):
  - Hueytown, Alabama
  - Chandler, Arizona
  - Sierra Vista, Arizona
  - Tucson, Arizona
  - Sherman, Arkansas
  - Sherwood, Arkansas
  - Carmichael, California
  - Garden Grove, California
  - Laguna Hills, California
  - Long Beach, California
  - Paramount, California
  - Rancho Cucamonga, California
  - Roseville, California
  - Sacramento, California
  - San Diego, California
  - San Ramon, California
  - Tustin, California
  - Westlake Village, California
  - Bristol, Connecticut
  - Boynton Beach, Florida
  - Hialeah, Florida
  - New Smyrna Beach, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Conyers, Georgia
  - Newnan, Georgia
  - Stockbridge, Georgia
  - Rockford, Illinois
  - Metairie, Louisiana
  - Prince Frederick, Maryland
  - Stevensville, Michigan
  - Olive Branch, Mississippi
  - Egg Harbor, New Jersey
  - Albuquerque, New Mexico
  - Rochester, New York
  - Wilmington, North Carolina
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Yukon, Oklahoma
  - Portland, Oregon
  - Lansdale, Pennsylvania
  - Salisbury, South Carolina
  - Chattanooga, Tennessee
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - South Ogden, Utah
  - Chesapeake, Virginia
  - Norfolk, Virginia
  - Lakewood, Washington

REFERENCES:
- [Derived] Fass R, Inadomi J, Han C, Mody R, O'Neil J, Perez MC. Maintenance of heartburn relief after step-down from twice-daily proton pump inhibitor to once-daily dexlansoprazole modified release. Clin Gastroenterol Hepatol. 2012 Mar;10(3):247-53. doi: 10.1016/j.cgh.2011.11.021. Epub 2011 Dec 7. PMID 22155561
- See also: Dexilant Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=9efb34b3-fb69-4190-a2be-a90b8cb94e25&filetypecode=DEXILANTPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 45 investigative sites in the United States from 10 February 2009 to 15 April 2010.
Pre-assignment Details: Participants with a diagnosis of gastroesophageal reflux disease, whose symptoms were well controlled on twice daily proton pump inhibitors, were enrolled in the study and received a once-daily (QD) dexlansoprazole modified release (MR) capsule in the morning and a matched placebo capsule in the evening.
Period: Overall Study
Arm/Group | Dexlansoprazole MR QD
Started | 178
Completed | 163
Not Completed | 15
Not completed — Adverse Event | 7
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Participant Reported Lack of Efficacy | 1
Not completed — Participant Took Excluded Medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 178
Age, Customized [Number; unit: participants]
  <45 years | 56
  45 to <65 years | 94
  ≥65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 71

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Remain Well Controlled After Switching From Their Current Twice-daily Proton Pump Inhibitor Therapy to Dexlansoprazole MR.
Description: Well-controlled participants were defined to be participants who completed the study having at least 23 days of evaluable diary entries between Days 15 and 42, inclusive, and had ≤4 occurrences of heartburn during this period.
Time Frame: Week 3 through Week 6
Population: Values are from the Full Analysis Set.
Measure: Number; unit: percent of participants
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 142
percent of participants | 88

2. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOL) - Daily Activities Subscale in Participants Who Remain Well-controlled.
Description: PAGI-QOL is a 30-item self-reported instrument assessing health-related quality of life impact of upper gastrointestinal disorders. It includes 30 items across five subscales (daily activities, clothing, diet/food habits, relationship, psychological well-being and distress), scored on a 6-point Likert scale with subscale and total score ranging from 0 (none) to 5 (all the time). For reporting purposes, the scores are reversed and higher scores reflect improved quality of life and positive changes from baseline indicate improved quality of life.
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.05 (0.467)

3. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOL) - Clothing Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 2
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.02 (0.717)

4. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOL) - Diet and Food Habits Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 2
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.27 (0.858)

5. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOL) - Relationship Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 2
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.10 (0.415)

6. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOL) - Psychological Well-being Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 2
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.03 (0.541)

7. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders - Quality of Life (PAGI-QOL) - Total Score in Participants Who Remain Well-controlled.
Description: as for outcome 2
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.09 (0.417)

8. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Nausea/Vomiting Subscale in Participants Who Remain Well-controlled.
Description: PAGI-SYM is a 20-item self-reported questionnaire that measures symptom severity of upper gastrointestinal disorders across six subscales (nausea/vomiting, fullness/early satiety, bloating, upper abdominal pain, lower abdominal pain, heartburn/regurgitation) which are summarized by individual subscale scores and a total score. The items are rated on a 6-point Likert scale with subscale and total score ranging from 0 (none) to 5 (very severe). Higher scores indicate higher symptom severity and thus negative changes from baseline indicate decrease in symptom severity.
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | 0.00 (0.522)

9. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Fullness/Early Satiety Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 8
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | -0.10 (0.730)

10. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Bloating Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 8
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | -0.20 (1.024)

11. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Upper Abdominal Pain Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 8
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | -0.08 (0.981)

12. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Lower Abdominal Pain Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 8
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | -0.03 (0.628)

13. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Heartburn/Regurgitation Subscale in Participants Who Remain Well-controlled.
Description: as for outcome 8
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | -0.14 (0.729)

14. Secondary Outcome: Change From Baseline in Patient Assessment of Upper Gastrointestinal Disorders - Symptom Severity Index (PAGI-SYM) - Total Score in Participants Who Remain Well-controlled.
Description: as for outcome 8
Time Frame: Baseline and Week 6.
Population: Values are from the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexlansoprazole MR QD
Number analyzed (Participants) | 120
units on a scale | -0.09 (0.563)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after the last dose of single-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole MR QD
Serious Adverse Events (participants affected / at risk) | 6/178
Other Adverse Events (participants affected / at risk) | 34/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole MR QD (N=178)
Diverticular perforation (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Suicidal behaviour (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole MR QD (N=178)
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 5
Nasopharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 5
Headache (Nervous system disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.